CLINICAL TRIAL: NCT01297088
Title: Open-label, Single Center Study of the 18F-labeled PET/CT (Positron Emission Tomography / Computed Tomography) Tracer BAY86-9596 Following a Single Intravenous Administration of 300 MBq (Corresponding to ≤ 18 µg Mass Dose) for Evaluation of Biodistribution in Pathological Tissue in Patients With Cancer or Inflammation
Brief Title: PET/CT (Positron Emission Tomography / Computed Tomography) Investigations With BAY86-9596 (18F) (300 MBq) Following Single Intravenous Administration in Patients With Cancer or Inflammations.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Life Molecular Imaging SA (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 15146
Record Dates: First submitted 2011-02-14; First posted 2011-02-16 (Estimated); Last update posted 2013-01-21 (Estimated); Status verified 2013-01

CONDITIONS: Diagnostic Imaging
Keywords: Proof of Mechanism; Phase I; Neoplasm; Inflammation
MeSH Terms: conditions — Neoplasms; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: BAY86-9596

INTERVENTIONS:
Drug: BAY86-9596 — One single dose administration of a diagnostic agent

SUMMARY:
The study will be conducted as an open label, single-center, single dose and biodistribution study in patients with cancer or inflammation. 56 patients will be selected among the patients undergoing the screening examination conducted within 3 weeks before drug administration. Single dose of the study drug will be administrated in a dose of 300 MBq to these patients. The follow-up period contains the end-of-study telephone interview 5-8 days following the treatment. Key measurements are the PET/CT image acquisitions within a time frame of about 2 hours after the single injection of BAY86-9596.

ELIGIBILITY:
Inclusion Criteria:

* Cancer Patients

  * Patient had an Fluorodeoxyglucose (FDG) Positron Emission Tomography (PET)/Computer tomography(CT) performed 14 days prior to treatment with BAY86-9596 for detection, or staging, or restaging, or therapy response assessment that still showed tumor mass with high certainty, for cancers such as

    * Colorectal cancer,
    * Breast cancer (female patients),
    * Hepatocellular carcinoma (HCC) and the cancers under colorectal cancer to hepatocellular carcinoma (HCC) are histologically confirmed (Exception, based on diagnostic criteria for the management of hepatocellular carcinoma: Histological diagnosis of hepatocelluar carcinoma is not necessary if the nodule is larger than 2 cm, has been visualized in two dynamic imaging studies and shows arterial hyperenhancement and washes out in the venous phase.)
  * Patient has prostate cancer (primary or recurrent), still shows tumor mass (primary tumor and/or lymph node metastasis and/or distant metastasis) and the primary cancer disease is histologically confirmed
  * Patient has brain metastasis (strong evidence from imaging modalities), and the primary cancer disease is histologically confirmed.
  * Patient has a primary malignant brain tumor which is either confirmed by histology, or a positive cytology of cerebrospinal fluid, or imaging modalities (such as MRI, CT) strongly support the diagnosis of brain tumor.
  * Patient has some other cancer (such as ovarian cancer, melanoma), preferably with an FDG PET/CT available, and the primary cancer is histologically confirmed.
* Inflammation Patients

  * Patient with inflammatory disease having inflammatory focus/foci. An FDG PET/CT of the inflammation is available.
  * Patient underwent FDG PET/CT during the inflammation. The maximum interval between FDG PET/CT and examination with BAY86-9596 is 5 days, performance of both examinations on two subsequent days is recommended.

Exclusion Criteria:

* Concurrent severe and/or uncontrolled and/or unstable medical disease other than cancer or inflammation (e.g. poorly controlled diabetes, congestive heart failure, myocardial infarction within 12 months prior to planned injection of BAY86-9596, unstable and uncontrolled hypertension, severe pulmonary disease, chronic renal or hepatic disease which could compromise participation in the study. When considering hepatic function in hepatocellular cancer patients, the Child-Pugh score is applied, a score > 7 will be considered an exclusion criterion.
* Known sensitivity to the study drug or components of the preparation
* Drug abuse/dependence or history of recovered alcohol dependence.
* Patient has completed participation in another clinical study involving administration of an investigational drug in the preceding 4 weeks or is participating in any other clinical trial during this study
* Previous participation in treatment phase in this study
* Unwillingness or inability to comply with the protocol
* Patient fulfils criteria which in the opinion of the investigator preclude participation for scientific reasons, for reasons of compliance, or for reasons of the patient's safety.
* Patients with inflammatory disease with known tumor where images of tumor lesions may overlap with inflammatory lesions, or tumor patients with known inflammatory diseases (e.g. autoimmune diseases), where images of inflammatory lesions may overlap with tumor lesions.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-05; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
BAY86-9596 lesion detection rate (overall number of lesions identified). | up to 2 hours
Overall image quality (poor, satisfactory, excellent; based on investigator's experience with 18F-labeled PET tracers) | up to 2 hours
BAY86-9596 accumulation score in identified lesions (low accumulation, high accumulation). | up to 2 hours
Comparative score BAY86-9596 versus FDG. If an FDG PET/CT is not available (in malignant brain tumors or in brain metastasis), this comparison will be done with routine imaging modalities such as CT or MRI, or choline PET/CT. | up to 2 hours
Comparison of BAY86-9596 accumulation with lesions identified in histology of prostate cancer. | up to 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Singapore, Singapore